CLINICAL TRIAL: NCT06954701
Title: Evaluation of a Novel Personalizable Pessary for the Treatment of Pelvic Organ Prolapse
Brief Title: Evaluation of a Personalizable Pessary for Pelvic Organ Prolapse
Acronym: NPP-POP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Cosm Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00149345
Record Dates: First submitted 2025-04-17; First posted 2025-05-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Organ Prolapse (POP)
Keywords: Pelvic Organ Prolapse; Pessary
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Non-Inferiority study. Patients will act as their own controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Novel Personalizable Pessary Arm (Other): All patients in the study have previously been fit and used a standard pessary prior to the trial. They will use their standard pessary for one month. All participants will then be fit with a novel pessary, which they will use for 3 months.
  Interventions: Device: Novel Personalizable Pessary

INTERVENTIONS:
Device: Novel Personalizable Pessary — Novel personalizable pessary.

SUMMARY:
Pelvic organ prolapse (POP) is a common health issue. It will impact about half of Canadian women over their lifetime. With POP, organs like the bladder, uterus, and bowel may push into the vagina. Women may experience urine leakage, physical discomfort, and embarrassment. Aside from surgery, a common treatment for POP is the use of pessaries. Pessaries are removable devices placed inside the vagina that can relieve POP symptoms. Unfortunately, pessaries have fixed sizes and three in ten patients cannot find the right fit. Pessaries can cause bleeding and discomfort if they do not fit well or are not removed and cleaned regularly. Almost half of patients who wear pessaries stop using them because of these issues. There is a need for a better pessary treatment for patients.

The investigators have developed a new pessary that has the natural shape of the vagina. This pessary is easier to remove and re-insert. The pessary is also custom fit for each patient. In this study, the investigators will compare our new pessary to traditional pessaries. Study participants who have been fit with a traditional pessary will be asked to use our new pessary design for 3 months. Study participants will fill out questionnaires about their POP symptoms. The investigators will also ask patients to provide their feedback on comfort and how easy it is to use the new pessary. This study could open up new possibilities for treating POP across Canada and around the world.

DETAILED DESCRIPTION:
Purpose: Pelvic organ prolapse (POP) impacts 50% of Canadian women in their lifetime. POP can be associated with voiding dysfunction, bowel dysfunction, and sexual dysfunction, thereby impacting quality of life. Pessaries are insertable devices used to conservatively manage POP, avoiding surgery. While surgery is effective for managing POP is effective in the short term, recurrence is common and occurs in at least 30% of patients. Traditional pessaries have not undergone any design changes in the last 50 years, and up to 30% of patients can not find a pessary that fits them well. Of the patients who do find a well fitting pessary, not all patients are independent with pessary care and up to 50% will discontinue their use in the first year either due to this lack of independence with care or due to complications associated with their use. With the advent of 3D printing technology, the possibility for a personalizable and easier to use design has become a reality. The investigators have designed a novel personalizable pessary (NPP) to address the shortcomings of traditional vaginal pessaries.

Hypothesis: The NPP will be non-inferior to standard pessaries with regards to efficacy and safety.

Null Hypothesis: The mean difference score (μ study pessary-control) between baseline and study pessary on the Pelvic Floor Distress Inventory 20 (PFDI-20) is greater than 18.3, the upper equivalence limit, or lower than -18.3, the lower equivalence limit.

Justification: Pelvic organ prolapse (POP) is the descent of pelvic organs into the vagina. It is an overlooked, stigmatized, and growing women's health issue, affecting up to 50% of Canadian women. POP contributes to other pelvic floor disorders such as urinary and/or fecal incontinence, and sexual dysfunction. POP significantly affects mental health, contributing to diminished quality of life (QoL), social isolation, and increased risks of depression and anxiety. The prevalence and burden of POP are growing rapidly, tied to the growth of our aging population.

POP treatment encompasses surgical and non-surgical options. While surgery proves effective, POP recurrence rates are up to 70% within 5 years, requiring reoperation and increasing surgical complications to patients and imposing a substantial economic burden on healthcare. Moreover, wait times for POP surgery in Canada are increasing up to 50%, which further exacerbates the challenges faced by women in need of care. Vaginal pessaries are a non-surgical option to treat POP that can be very effective and are offered as first-line therapy by 75% of physicians. However, pessaries have several limitations. These include a trial-and-error fitting process, an inability to find the right fit for all patients, and difficulty in self-care (i.e., remove, clean, and reinsert). These issues can lead to complications and high discontinuation rates (up to 53% in one year). This underscores a significant predicament for patients grappling with the inability to secure an optimal pessary fit, compelling them to resort to surgery - an undesirable outcome despite the prevalent preference for non-surgical alternatives.

While pessaries have not undergone many changes over the last half century, recent advancements in 3D printing for medical applications offer an unprecedented level of control over structure geometry. Recently, initiatives to innovate personalized pessaries through 3D printing have begun by our team and others and are increasingly garnering attention. A recent editorial in the journal Urogynecology issued a "call to action" for "disruptive innovations" in pessaries to better serve this overlooked patient population. There is a significant unmet need for improved pessary treatment options to ensure inclusive non-surgical care for patients with POP.

To address the critical gap in POP treatment in the current paradigm, our team has developed a novel expansible personalized pessary by leveraging 3D printing, enabling the development of more complex shapes. This novel pessary design, inspired by the anatomical shape of the vagina, addresses challenges related to the fitting process, finding the optimal fit, performing self-care, and ultimately improving the QoL for women experiencing POP. The objective of this research is to evaluate the safety and efficacy of this novel pessary in treating the symptoms of POP in patients impacted by this condition. optimize the design of this novel pessary and demonstrate its feasibility in patients with POP. Success of this research could unlock the potential for an improved non-surgical treatment option for POP, the impact of which extends beyond Canada, offering a global impact on the well-being of women.

The study pessary is made of biocompatible silicone similar to commercially available pessaries. The material and production processes are identical to Cosm Medical's Gynethotics Pessaries, currently approved by Health Canada (Medical Device License 110149) and available on the market.

Objectives: To assess the safety and efficacy of the NPP compared to traditional pessaries. Additional areas of assessment include proportion of patients able to be fit with the NPP and proportion of patients able to self-manage use of the NPP.

Research Method/Procedures: This is a single site, prospective, open label, non-inferiority study of a medical device. This study focuses on optimizing the sizing and personalization of the NPP using physical assessment and provides an opportunity to optimize the design for improved outcomes through patient and provider feedback. Study participants will act as their own controls. Forty-three patients with varying pessary histories will be recruited. The study participants will use a standard pessary for one month. Participants will then use the NPP for 3 months. The primary endpoint is the change in PFDI-20 score when comparing the participant's use of a standard pessary, as well as a comparison of prevalence and severity of adverse events. Secondary outcomes include changes in patient-reported symptoms, sexual function, and quality of life, as well as visual analogue score ratings on ease of NPP insertion/removal and comfort. Application to Health Canada of the NPP is pending.

Plan for Data Analysis: Data will be analysed with the assistance of a statistician. The primary outcome, assessed by PFDI-20 scores, will be reported as means and standard deviations or medians and interquartile ranges (IQR), based on the normality of the distribution. Scores will be matched and compared between the traditional and study pessary devices. In instances where the distribution is normal, a two-tailed matched t-test will be utilized; conversely, the Wilcoxon Signed-Rank Test will be implemented for non-normal distributions. Furthermore, to evaluate adverse events between matched groups, McNemar's Test will be employed. Sensitivity analyses will be conducted as exploratory analyses to compare outcomes across intention-to-treat (ITT), per protocol, and as-treated subgroups.

As success criterion for the analysis, Wiegersma et al identified the minimal important change for the PFDI-20 in women opting for conservative management of prolapse as 13.5-18.3 points. The investigators will conduct two one-sample equivalence t-tests, each with an alpha of .05, to test the composite null hypothesis that the mean difference score (μStudyPessary-control) between baseline (current pessary) and study pessary is either greater than 18.3 or less than -18.3:

The investigators will reject the null hypothesis if the maximum p-value from both tests is less than 0.05.

All continuous variables will be described using means and standard deviations or medians and interquartile ranges as appropriate. For categorical variables, frequencies and percentages will be reported. Specific assessments include the Pelvic Floor Impact Questionnaire Short Form 7, Pelvic Organ Prolapse / Urinary Incontinence Sexual Questionnaire (International Urogynecological Association Revised), and objective assessments of ability to support prolapse, all treated as continuous variables. Pain associated with insertion and removal will be assessed using Visual Analog Scale scores. Success and ease of fitting, as well as ease of insertion and removal, will be categorized, while the frequency of self-management will be reported as a count or numeric variable.

ELIGIBILITY:
Inclusion Criteria:

* Patients assigned female at birth
* At least 18 years old at time of screening
* Patients with symptomatic POP using a pessary for ≥ 3 months
* Capable of giving informed consent
* Fluency in English

Exclusion Criteria:

* Pregnancy
* Short vaginal length (total vaginal length <5 cm) or subjective vaginal narrowing
* Vaginal erosion due to current pessary
* Presence of vesicovaginal fistula
* Presence of rectovaginal fistula
* Current treatment for vaginal, rectal, or bladder tumor
* Presence of open wound or tear near vagina or anus by exam prior to removal of current pessary
* Presence of pelvic, vaginal, or urinary infection requiring treatment
* Ongoing treatment of recurrent urinary tract or vaginal infections
* Inflammatory bowel disease
* Chronic pain syndromes of pelvic or anorectal origin
* Previous pelvic floor surgery in last 12 months
* Congenital malformation of bladder, rectum, or vagina
* Significant medical condition interfering with study participation (psychologic, neurologic, active drug/alcohol abuse, ambulatory restrictions, etc.)
* Planning pregnancy in next 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Pelvic Floor Distress Inventory-20 (PFDI-20) score | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Comparison of PFDI-20 scores between standard pessary and the study device. Score range 0-300, with higher scores indicating greater burden of pelvic floor symptoms.

SECONDARY OUTCOMES:
Change in Pelvic Floor Impact Questionnaire (PFIQ-7) | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Comparison of PFIQ-7 scores between standard pessary to the study device. Scoring ranges from 0-300, with higher scores indicating increasing burden of symptoms.
Change in Patient Global Impression of Improvement (PGI-I) | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Change in PGI-I between standard pessary and study device. Utilized to assess symptoms of stress urinary incontinence. Scored from 1 (symptoms very much better) to 7 (symptoms very much worse).
Change in the subscale Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6). | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Change in the POPDI-6 subscale within the PFDI-20 between standard pessary and study device. Scoring ranges from 0-100, with higher scores indicating increasing burden of symptoms.
Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, International Urogynecologic Association-Revised (PISQ-IR) | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Change in PISQ-IR score between standard pessary and the study device. Scoring ranges from 0-300, with higher scores indicating increasing burden of symptoms.
Quality of life (QoL) questionnaire, i.e., the European-Quality of Life-5 Dimensions - 5 Levels (EQ-5D-5L) | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Change in EQ-5D-5L score between standard pessary and the study device. Scores from this tool range from 1 to 5, with higher numbers reflecting more severe problems, and are used to assess the areas of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Objective Pelvic Organ Prolapse - Quantification (POP-Q) Assessment | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Comparison of points Ba and Bp in the POP-Q system between standard pessary and study device. Measurements on the POP-Q reflect objective measurements in centimetres of a patient's prolapse.
Visual Analogue Score (VAS) - Global Satisfaction | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Comparison of global satisfaction between standard pessary and the study device using VAS. Measure from 0 to 100 with lower numbers representing lower satisfaction.
Visual Analogue Score (VAS) for Ease of Pessary Insertion | From enrolment to end of treatment.
  Comparison of VAS scores assessing ease of pessary insertion by study participants between standard pessary and study device. Scored from 0 to 100 with higher numbers reflecting easier pessary insertion.
Visual Analogue Score (VAS) for Self-Management | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Comparison of VAS scores assessing self-management by study participants between standard pessary and study device. Score from 0 to 100 with higher scores indicating higher ability for patient self-management of the study device.
Visual Analogue Score (VAS) - Pain with Insertion | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Comparison of VAS scores assessing pain associated with pessary insertion by study participants between standard pessary and study device. Scores from 0 to 100 with higher scores indicating higher levels of patient reported pain with pessary insertion.
Visual Analogue Score (VAS) - Pain with Device Removal | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Comparison of VAS scores assessing pain with pessary removal by study participants between standard pessary and study device. Scores from 0 to 100 with higher scores indicating higher levels of patient reported pain with pessary removal.
Adherence | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Assessment of patient self-reported adherence to treatment with standard pessary and study device.

OTHER OUTCOMES:
Study Pessary Fit | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Proportion of subjects successfully fit with the study pessary
Patient Self-Management | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Percentage of patients able to self-manage the study pessary (self-reported).
Change in frequency of pessary removal for self-managers | Approximately 4 months (1 month of standard pessary use and 3 months of study device use).
  Assessment by self-report of frequency of pessary insertion/removal if independent with pessary care.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Vasas, MD, Study Director — University of Alberta
Locations (1):
- Dale Sheard Centre for Solutions in Women's Health, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No